CLINICAL TRIAL: NCT03951090
Title: Geriatric Assessment Reporting in Real Time (GARRT) in Non-electively Hospitalized Older Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 1538
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an un-blinded, 2-arm randomized control trial of a brief, user friendly GA report in real time which summarizes GA-identified deficits and includes recommendations for evidence informed multidisciplinary interventions to address these deficits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GARRT Arm (Experimental): Participants in this arm complete an brief geriatric assessment, and the results of these assessments are given to providers with recommendations to address deficits identified by the geriatric assessment
  Interventions: Other: Results of the brief geriatric assessment
- Control Arm (Active Comparator): Providers of participants of this group will not receive the results of the brief geriatric assessments. These participants will receive standard of care treatment
  Interventions: Other: No results of brief geriatric assessments

INTERVENTIONS:
Other: Results of the brief geriatric assessment — Providers will receive results of the brief geriatric assessment with recommendations for address deficits identified through the results of the brief geriatric assessment
  Arms: GARRT Arm
Other: No results of brief geriatric assessments — Providers will not receive results of the brief geriatric assessment. Participants will receive standard of care treatment
  Arms: Control Arm

SUMMARY:
This study prospectively evaluates the impact of geriatric assessment reporting in real-time (GARRT) on key hospital based outcomes in a cohort of non-electively hospitalized older (> 70 years) adults with cancer.

DETAILED DESCRIPTION:
This study evaluates the impact of geriatric assessment reporting in real-time (GARRT) on key hospital based outcomes in non-electively hospitalized older (> 70 years) adults with cancer. Participants will be randomly assigned to the GARRT group, or the control group. All participants will fill out user friendly questionnaire called the geriatric assessment. The results of the geriatric assessment will be given to the physicians of participants in the GARRT group in real-time. The physicians of participants in the control group will not receive real time results.

This study will compare the referral rates of participants in each group to determine if providing real-time results of the geriatric assessment impact referral rates.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older.
* English speaking.
* Admitted to UNC Hospitals non-electively within 72 hours.
* Biopsy proven solid tumor or myeloma or lymphoma.
* Newly diagnosed cancer patients for whom active cancer directed therapy is planned within the next six months or patients on active cancer directed therapy either currently or within the previous 6 months.
* Signed written IRB-approved informed consent.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria at baseline will be excluded from study participation. Patients with a life expectancy <6 weeks
* Patients who are <48 hours post-surgery.
* Patients who are admitted to an intensive care setting.
* Patients with acute myeloma lymphoma (AML) or other high grade hematologic malignancies.
* Patients undergoing bone marrow transplant or admitted to the bone marrow transplant unit.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Referral rate for GA-identified deficits in intervention and control groups | 2 years
  Number of participants with at least one referral for a GA-idenfied deficit

SECONDARY OUTCOMES:
Referral to Physical and Occupational therapy | 2 years
  Number of times physical and occupation therapy referral was given in Intervention and Control group
Referral to Geriatic Consultation | 2 years
  Number of times a Geriatric Consultation referral was given in Intervention and Control group
Referral to Clinical Pharmacist | 2 years
  Number of times Clinical Pharmacist referral was given in Intervention and Control group
Referral to Nutritionist | 2 years
  Number of times Nutritionist referral was given in Intervention and Control group
Referral to psyhcosocial support team | 2 years
  Number of times psychosocial support referral was given in Intervention and Control group
Physician Reported New information | 2 years
  Number of times physicians answer "yes" to the questions "did report provide new information about patient deficits that would warrant a referral"
Physician Reported Satisfaction | 2 years
  Number of times physician indicate "yes" report was helpful when asked "Is this report useful"

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Jolly, MBBS, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States